CLINICAL TRIAL: NCT02917785
Title: Testing the Efficiency of Karman Curette in the Treatment of Misoprostol Failure in Women With Missed Abortion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 177-16-MMC
Record Dates: First submitted 2016-09-07; First posted 2016-09-28 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-09

CONDITIONS: Abortion, Missed
MeSH Terms: conditions — Abortion, Missed

ARMS (2):
- Karman curettage (Experimental): after a retained product of interception is observed in ultrasound examination, the women in this arm will undergo Karman curretage.
  Interventions: Device: Karman curettage
- Control (No Intervention)

INTERVENTIONS:
Device: Karman curettage
  Arms: Karman curettage

SUMMARY:
the purpose of this study is to examine the success rates of Karman curettage in completing the abortion after failed recurred treatment with Misoprostol for women with missed abortion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women diagnosed with missed abortion treated in Meir Medical Center.
* The abortion occured during the first trimester of pregnancy.
* Patients who chose drug therapy (Misoprostol), after retained products of conception were evident on ultrasound.

Exclusion Criteria:

* patients with mullarian abnormality (i.e. septal uterus, myoma etc.)
* patients with significant bleeding
* Endometrial wall (residua) greater than 20 mm.
* known or suspected infection
* known clotting defect
* women after cesarean section
* closed cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Completing the abortion | 1 month
  completing the abortion until the scheduled day for hysteroscopy, thus preventing the need for hysteroscopy

SECONDARY OUTCOMES:
number of days of bleeding | 3 months
  asking the patient how many days of bleeding did she have after the procedure
pregnancy | 3 months
  asking the patient if she is currently pregnant
Pain intensity | 3 months
  asking the patient about the intensity of the pain during and after the procedure, as measured with NRS-11 pain scale
infection | 3 months
  asking the patient if she was diagnosed with any infection signs
number of sick days | 3 months
  asking the patients how many sick leave days did she take
number of days of abstinence from sexual intercourse | 3 months
  asking the patient how many days did she abstain from sexual intercourse after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Meir Pomeranz, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical center, Kfar Saba, Israel

REFERENCES:
- [Derived] Pomeranz M, Goren Gepstein N, Ovadia M, Klein Z, Daykan Y, Schonman R, Arbib N. A novel method for office aspiration curettage in cases of retained products of conception: A randomized controlled trial. Acta Obstet Gynecol Scand. 2021 Nov;100(11):2076-2081. doi: 10.1111/aogs.14245. Epub 2021 Aug 31. PMID 34467531